CLINICAL TRIAL: NCT03655470
Title: Screening and Brief Intervention for Suicidality and Nonsuicidal Self-Injury Among Youth in the Juvenile Justice System
Brief Title: Safety Planning in Juvenile Justice for Suicidal Youth
Acronym: Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1804002013; 1R34MH114307-01A1 (NIH)
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Suicidal Ideation; Suicide, Attempted; Nonsuicidal Self-injury
Keywords: suicidal behavior; nonsuicidal self injury; adolescents
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2 group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind; participants will not be told to what condition they are assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Planning (Experimental): This brief intervention, consists of an in-person and follow-up phone call that are based on cognitive behavioral principles designed to help identify a concrete list of coping strategies and social supports that youth can utilize preceding or during a crisis to lower imminent risk of nonsuicidal self-injury or suicidal behavior.
  Interventions: Behavioral: Safety Planning
- Standard Care (Active Comparator): If a teen has a positive screen for suicide risk, the Probation Officer completes a "secondary screener" built into the court screening instrument to determine whether there is concern of current and/or imminent risk. If a teen endorses nonsuicidal self-injury more than once in the prior year, then the Probation Officer asks about frequency and severity. If there is ongoing concern of risk for self-injurious behavior, then the Probation Officer arranges for a crisis evaluation in the Emergency Department. If the teen is not judged to be at imminent risk, the Probation Officer makes a referral back to the current treatment provider or to a community mental health clinic. In either case, the parents and youth receive a packet with mental health resources
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Safety Planning — Safety planning is an individual coping intervention to reduce suicidal risk in adolescents
  Arms: Safety Planning
Behavioral: Standard care — Standard care entails sending an adolescent for an emergency evaluation for suicidal risk in an Emergency Department
  Arms: Standard Care

SUMMARY:
This study will examine the feasibility and acceptability of a program designed to conduct safety planning with youth in the juvenile justice system who are at risk for a suicide attempt and/or self-injury and to increase the possibility of them receiving outpatient mental health treatment. After training staff in the intervention, the investigators will pilot test the safety planning intervention and gather information on how well it worked on reducing self-harm, getting families to follow up with referrals for mental health care, and how often they attend treatment.

DETAILED DESCRIPTION:
The Juvenile Justice System (JJS) has not implemented any evidenced-based interventions that address suicidal behavior or nonsuicidal self-injury, hereafter referred collectively to as self-injury, with JJS-involved youth. This application proposes to test a scalable intervention, safety planning, that aims to reduce self-injury in adolescents involved in the JJS. Safety planning, which can be a stand-alone brief intervention, was cited as a best practice by the Suicide Prevention Resource Center/American Foundation for Suicide Prevention Best Practices Registry for Suicide Prevention. This study will have two phases. In Phase I, the investigators will conduct an open trial with 10 adolescents which will allow us to make any modifications necessary for using the protocol in a Probation Department. The investigators will then randomize 60 youth on Probation who screen positive for recent self-injury into standard care or the safety planning intervention. Counselors with community mental health experience embedded in Probation will conduct the intervention, consistent with the co-responder model found across JJS in the U.S. in which a Probation Officer works collaboratively with a mental health professional to coordinate care. In order to further conduct the study under conditions most relevant to a future implementation trial, the investigators will also employ a training approach that has been successfully implemented in a psychiatric hospital with Bachelors and Masters level staff. In Phase II, of the study, the investigators will: a) conduct qualitative interviews in Probation about attitudes toward the intervention as well as barriers to a future, larger implementation trial; and b) contract with the National Center for Mental Health and Juvenile Justice to conduct a Sequential Intercept Model (SIM) Mapping. The SIM is a conceptual framework to outline a series of "points of interception" along the JJS continuum in a state where screening and brief intervention may be implemented. In the Mapping, the investigators will examine the JJS continuum from arrest; to an initial hearing; to jail awaiting trial or adjudication; incarceration; to release or reentry; and finally, to community supervision. These data will provide a working framework to help assess current views within the statewide JJS as a starting point to proposing a future, larger trial. This research also has the potential to directly inform treatment practices in JJ settings and has significant implications for scalability and dissemination in order to build a stronger, more effective system of mental health/JJS collaboration around self-injury screening and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardian available to consent for juvenile's participation
* Juvenile and parents are English or Spanish speaking
* Juvenile flags in on the screening measure used in court with respect to suicidal ideation or nonsuicidal self-injury.

Exclusion Criteria:

* None

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown U
Locations (2):
- United States (2):
  - Rhode Island Family Court, Providence, Rhode Island
  - Brown Univerity, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The final study protocol will contain the information necessary to reproduce the findings in other populations. The protocol will include a copy of this grant application including Specific Aims and study population; recruitment and enrollment information; the measures collected and coding of the measures and subscales; the clinician intervention procedures; data analyses; syntax for data summary, and data analysis plans
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of all follow-up data
Access Criteria: Contact PI

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Safety Planning | Standard Care
Started | 29 | 30
Completed | 23 | 23
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Planning | Standard Care | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.75 (1.35) | 15.07 (1.58) | 14.93 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 16 | 22 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 19 | 22 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 12 | 15 | 27
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59
Massachusetts Youth Screening Instrument - Angry/Irritable subscale, [Mean (Standard Deviation); unit: units on a scale] — MAYSI subscale range 0 - 9, higher indicates higher levels of anger and irritability
  units on a scale | 4.21 (2.90) | 4.73 (3.07) | 4.47 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: Change in Suicidal Ideation
Description: Score on Suicidal Ideation Questionnaire; higher is worse; range 0 to180
Time Frame: Past month ideation at 1 and 3 month follow-up points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety Planning | Standard Care
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline SIQ | 8.90 (12.19) | 8.97 (14.37)
  1-month follow-up | 12.27 (17.57) | 7.36 (15.54)
  3-month follow-up | 10.15 (14.81) | 4.54 (7.38)
Statistical Analysis 1: Comparison: Safety Planning vs Standard Care; Test type: Superiority; p = .30, Mixed Models Analysis; Mean Difference (Final Values) = .59, Standard Error of Mean .07

2. Secondary Outcome: Suicide Attempts
Description: Whether a participant reported a suicide attempt
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Planning | Standard Care
Number analyzed (Participants) | 29 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Safety Planning | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

LIMITATIONS AND CAVEATS:
The major limitations were: 1) identification of participants eligible for the study in the various sections of the juvenile legal system with different frontline staff; and 2) follow-up rate for enrolled participants was no as high as expected due primarily to the fact that most participants exited the juvenile legal system at 3 months and therefore, at times, were unwilling to complete follow-up because they were no longer in the family court system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03655470/Prot_SAP_001.pdf
  • Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03655470/ICF_000.pdf